CLINICAL TRIAL: NCT07376811
Title: Effect Of Sleeping Posture Guidance On Sleep Quality In Patients With Rotator Cuff Syndrome Undergoing Physical Therapy: A Randomized Clinical Trial
Brief Title: Effect Of Sleeping Posture Guidance On Sleep Quality In Patients With Rotator Cuff Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Unifesp Escola Paulista de Medicina (Unknown)
Responsible Party: Principal Investigator, Paulo Santoro Belangero, Affiliate Professor Of The Department Of Orthopedics And Traumatology Paulista Medical School / Federal University Of São Paulo (UNIFESP) Sports Medicine And Physical Activity Division, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 93319125.3.0000.5505
Record Dates: First submitted 2026-01-14; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Rotator Cuff Syndrome; Rotator Cuff Injury; Sleep Disorder (Disorder)
Keywords: rotator cuff syndrome; sleep quality; sleeping position; physical therapy; randomized controlled trial; shoulder pain; rehabilitation
MeSH Terms: conditions — Rotator Cuff Injuries; Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders; Shoulder Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: This is a two-arm, parallel-group randomized clinical trial designed to compare the efficacy of two conservative treatment approaches. Participants diagnosed with Rotator Cuff Syndrome (RCS) are randomly allocated to one of two groups: an Active Comparator group (Standard Physical Therapy) or an Experimental group (Standard Physical Therapy combined with Sleeping Posture Guidance). The study evaluates outcomes at three distinct time points: baseline (T0), immediate post-intervention at 5 weeks (T5), and a long-term follow-up at 12 weeks (T12).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Comparator group (Physical Therapy) (Active Comparator): Participants receive the same 5-week standard physical therapy protocol (10 sessions, twice weekly) including manual therapy and progressive exercises, following evidence-based clinical practice guidelines for Rotator Cuff Syndrome.
  Interventions: Procedure: Physical Therapy
- Experimental group (Physical Therapy combined with Sleeping Posture Guidance) (Experimental): Participants receive a 5-week standard physical therapy protocol (10 sessions, twice weekly) consisting of manual therapy and progressive exercises, plus structured education and guidance on sleeping positions and pillow use to optimize sleep quality.
  Interventions: Procedure: Physical Therapy; Behavioral: Physical Therapy + Sleep Guidance

INTERVENTIONS:
Procedure: Physical Therapy — This intervention is applied to all study participants (both groups). Participants receive the same 5-week standard physical therapy protocol (10 sessions, twice weekly) including manual therapy and progressive exercises, following evidence-based clinical practice guidelines for Rotator Cuff Syndrome.
Behavioral: Physical Therapy + Sleep Guidance — Participants receive structured education and guidance on sleeping positions and pillow use to optimize sleep quality.
  Arms: Experimental group (Physical Therapy combined with Sleeping Posture Guidance)

SUMMARY:
This study investigates sleep quality in patients with Rotator Cuff Syndrome (RCS) undergoing physical therapy treatment. Existing literature presents a gap regarding longitudinal studies evaluating the impact of physical therapy and different sleeping positions on sleep quality within this specific population. The central hypothesis is that physical therapy, combined with guidance on the best sleeping positions, reduces pain, improves shoulder function, and consequently promotes an improvement in sleep quality for RCS patients over time. The justification for this research lies in the need to better understand the relationship between physical therapy and sleep quality in RCS patients, aiming for the development of more effective and less invasive interventions. Previous studies have demonstrated that chronic pain, a common symptom of RCS, is intrinsically linked to sleep disturbances, which can lead to deleterious effects such as dopamine reduction, alterations in the descending pain modulation system, and central sensitization. Improvements in sleep quality have been observed after surgical procedures such as shoulder arthroscopy and arthroplasty, often associated with improved function and pain reduction. Thus, this study seeks to longitudinally evaluate whether physical therapy is capable of promoting a sustained improvement in sleep quality for patients with RCS

DETAILED DESCRIPTION:
Background and Rationale Rotator Cuff Syndrome (RCS) is a prevalent musculoskeletal condition characterized by pain and functional limitation, which significantly impacts patients' quality of life. While physical therapy is a standard conservative treatment for reducing pain and restoring shoulder function, its longitudinal effect on sleep quality remains under-researched. Chronic pain in RCS is intrinsically linked to sleep disturbances, potentially leading to central sensitization and alterations in the pain modulation system. This study aims to address the gap in literature regarding the added benefit of structured sleep posture guidance when combined with standard rehabilitation.

Study Design and Procedures This is a parallel-group, randomized controlled clinical trial with a 1:1 allocation ratio. The study is designed as a simple-blind trial, where the outcome assessors will be blinded to the participants' group assignments.

Participants will be recruited from a specialized orthopedic and physical therapy center. Following the initial assessment (T0), eligible participants will be randomly assigned to either the Control Group or the Intervention Group using a set of sealed, opaque envelopes generated by an independent researcher.

Intervention Protocols

Control Group (Standard Physical Therapy): Participants will undergo a standardized physical therapy protocol consisting of 10 sessions (twice weekly for 5 weeks). The sessions follow evidence-based clinical practice guidelines for RCS and include:

Education on ergonomics and modifications of activities of daily living. Articular mobilization and manual therapy techniques. Progressive resisted exercises, including both isometric and isotonic modalities, focused on analgesia and functional recovery.

Intervention Group (Physical Therapy + Sleep Posture Guidance): Participants in this group will receive the exact same 10-session physical therapy protocol as the Control Group. Additionally, they will receive structured and personalized sleep posture guidance during the first week, with monthly reinforcements. This additional intervention includes:

Specific instructions on ideal sleeping positions to minimize nocturnal shoulder stress (e.g., avoiding sleeping on the affected shoulder).

Practical guidance on the use of supportive pillows to maintain the shoulder in a neutral and comfortable position throughout the night.

Follow-up and Data Management The total duration of the active treatment phase is 5 weeks. Data collection occurs at three specific time points: baseline (Week 1), post-intervention (Week 5), and a late follow-up (Week 12). Assessments at Week 1 and Week 5 are conducted in person, while the Week 12 follow-up is conducted remotely via an online platform. Data will be stored and managed using secure digital platforms to ensure participant confidentiality and data integrity.

Statistical Plan Overview The sample size of 64 participants was calculated to detect significant changes in sleep quality based on established PSQI score variances from similar populations. Statistical analysis will utilize both descriptive and inferential methods, applying a significance level of p ≤ 0.05 with a 95% confidence interval. Univariate and bivariate analyses will be performed to examine the relationships between pain levels, shoulder function, and sleep quality over time.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and/or radiological diagnosis of Rotator Cuff Syndrome (RCS).
* Presence of shoulder pain for at least 3 months (chronic pain).
* Patients aged between 18 and 65 years.
* Patients referred for conservative physical therapy treatment.
* Ability to understand and answer the assessment questionnaires (PSQI, MSQ, ASES, and VAS).
* Voluntarily signing the Informed Consent Form (ICF).

Exclusion Criteria:

* History of surgical procedures on the affected shoulder.
* Presence of fractures or recent acute trauma in the shoulder or upper limb.
* Associated neurological disorders, inflammatory systemic diseases (e.g., Rheumatoid Arthritis), or adhesive capsulitis (frozen shoulder).
* Previous diagnosis of primary sleep disorders unrelated to pain (e.g., severe obstructive sleep apnea) already under clinical treatment.
* Recent history of corticosteroid injections in the shoulder (within the last 3 months).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in sleep quality between the Physical Therapy Group and the Physical Therapy + Sleeping Posture Guidance Group | Time Points: Baseline (Week 1), Post-intervention (Week 5), and Follow-up (Week 12)
  Change in Sleep Quality Score as Measured by the Pittsburgh Sleep Quality Index (PSQI)
  Description: The PSQI is a self-reported questionnaire that assesses sleep quality over a one-month interval. It consists of 19 individual items, creating seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
  Scoring: The global score ranges from 0 to 21, where lower scores indicate better sleep quality. A global PSQI score greater than 5 is considered an indicator of relevant sleep disturbances.
To compare the change in sleep quality between the Physical Therapy Group and the Physical Therapy + Sleeping Posture Guidance Group | Time Points: Baseline (Week 1), Post-intervention (Week 5), and Follow-up (Week 12).
  Change in Sleep Quality Score as Measured by the Pittsburgh Sleep Quality Index (PSQI)
  Description: The PSQI is a self-reported questionnaire that assesses sleep quality over a one-month interval. It consists of 19 individual items, creating seven "component" scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. The sum of scores for these seven components yields one global score.
  Scoring: The global score ranges from 0 to 21, where lower scores indicate better sleep quality. A global PSQI score greater than 5 is considered an indicator of relevant sleep disturbances.

SECONDARY OUTCOMES:
Change in Shoulder Function as Measured by the American Shoulder and Elbow Surgeons (ASES) Score | Baseline (Week 1), Post-intervention (Week 5), and Follow-up (Week 12).
  The ASES is a standardized assessment form used to evaluate shoulder function and pain. It consists of two sections: a patient self-evaluation and a clinical assessment. The patient section focuses on pain (measured by a Visual Analog Scale) and 10 items related to activities of daily living (e.g., dressing, grooming, and lifting objects).
  Scoring: The total score is converted to a 100-point scale, where 100 represents a normal, pain-free shoulder and 0 indicates severe disability and pain.
Change in Pain Intensity as Measured by the Visual Analog Scale (VAS) | Baseline (Week 1), Post-intervention (Week 5), and Follow-up (Week 12)
  The VAS (Escala Visual Analógica - EVA) is a unidimensional measure of pain intensity. It consists of a 10-centimeter line where the left end represents "no pain" (0) and the right end represents "the worst imaginable pain" (10). Patients are asked to mark the point on the line that best represents their current pain level.
  Scoring: The score is determined by measuring the distance (in centimeters or millimeters) from the "no pain" end to the patient's mark.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo S Belangero, PHD professor, Principal Investigator — Federal University of São Paulo
Locations (1):
- Instituto Buran, São Caetano do Sul, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hodgetts CJ, Leboeuf-Yde C, Beynon A, Walker BF. Shoulder pain prevalence by age and within occupational groups: a systematic review. Arch Physiother. 2021 Nov 4;11(1):24. doi: 10.1186/s40945-021-00119-w. PMID 34736540
- [Result] Cofield RH. Rotator cuff disease of the shoulder. J Bone Joint Surg Am. 1985 Jul;67(6):974-9. No abstract available. PMID 4019548
- [Result] Khazzam MS, Mulligan EP, Brunette-Christiansen M, Shirley Z. Sleep Quality in Patients With Rotator Cuff Disease. J Am Acad Orthop Surg. 2018 Mar 15;26(6):215-222. doi: 10.5435/JAAOS-D-16-00547. PMID 29517624
- [Result] Finan PH, Goodin BR, Smith MT. The association of sleep and pain: an update and a path forward. J Pain. 2013 Dec;14(12):1539-52. doi: 10.1016/j.jpain.2013.08.007. PMID 24290442
- [Result] Desmeules F, Roy JS, Lafrance S, Charron M, Dube MO, Dupuis F, Beneciuk JM, Grimes J, Kim HM, Lamontagne M, McCreesh K, Shanley E, Vukobrat T, Michener LA. Rotator Cuff Tendinopathy Diagnosis, Nonsurgical Medical Care, and Rehabilitation: A Clinical Practice Guideline. J Orthop Sports Phys Ther. 2025 Apr;55(4):235-274. doi: 10.2519/jospt.2025.13182. PMID 40165544
- See also: Survey link for participant data collection (Portuguese) — https://docs.google.com/forms/d/e/1FAIpQLSf_VU-3WfWQ6u7QgnDxoLi5E4K2FUNx86a4fJPB-drhc6g0uA/viewform

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT07376811/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-11): https://cdn.clinicaltrials.gov/large-docs/11/NCT07376811/ICF_001.pdf